CLINICAL TRIAL: NCT03263221
Title: Traumatic Proximal Femoral Fractures in Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Helmy, assistant lecturer, Assiut University
Other Study IDs: Proximal femoral fractures
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: reduction and fixation — Surgical procedures, as plating, Proximal Femoral Nail , Dynemic Hip screw and others procedures according to needed for each types

SUMMARY:
Statistical analysis for adult patients who were admitted to Assiut university hospital within one year with proximal femoral fractures.

Protocol of management include lines of treatment , hospital stay and results

DETAILED DESCRIPTION:
Case series prospective study All adult patients who were admitted to AUH with proximal femoral fractures within one year.

We will evaluate the real treatment protocol which was applied for those patients.

Surgical procedures, as plating, Proximal Femoral Nail , Dynemic Hip screw and others procedures according to needed for each types.

This epidemological study in proximal femoral fractures will provide an update on incidence, admission, hospital stay and surgical procedures. This information will assist health providers in planning hospital beds, surgical intervention, and risk prevention, moreover, this data can be use for farther clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* 1-Adult Age 2- Closed & Open fracture

Exclusion Criteria:

* 1- Childern 2-pathological fractures

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adults patients with proximal femoral fractures
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
• Statistical analysis for adult patients who were admitted to Assiut university hospital within one year with proximal femoral fractures | baseline
  This epidemological study in proximal femoral fractures will provide an update on incidence, admission, hospital stay and surgical procedures